CLINICAL TRIAL: NCT05319366
Title: Proteomics- og Metabolomics-undersøgelse af Materiale Ekstraheret Fra Ballonkatetre Anvendt Til Ballon-udvidelsesbehandling Hos Patienter Med Symptomatisk åreforkalkningssygdom
Brief Title: Atherosclerotic Lesion Proteomics by Harvesting Angioplasty Balloons (ALPHA).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Gorm Mork, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: H-21029011
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Angina, Stable; Angina, Unstable; Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); ST-segment Elevation Myocardial Infarction (STEMI); Vascular Diseases
Keywords: Proteomics; Metabolomics; Atherosclerosis; Angioplasty; Vascular surgery
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Vascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples from the baloon catherther or vascular surgery and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Stable angina: 50 patients with stable angina will be included and tissue samples from balloon cathether and blood samples will be collected
- Unstable angina/non-ST-segment elevation myocardial infarction: 50 patients with unstable angina/non-ST-segment elevation myocardial infarction will be included and tissue samples from balloon cathether and blood samples will be collected
- ST-segment elevation myocardial infarction: 50 patients with ST-segment elevation myocardial infarction will be included and tissue samples from balloon cathether and blood samples will be collected
- Controls: 50 patients without corornary arthery-related treatment will be included and tissue samples from balloon cathether and blood samples will be collected
- Vascular surgery: 25 patients who undergo will be included and tissue samples and blood samples will be collected

SUMMARY:
The purpose of the study is to identify proteins, metabolites and signal pathways related directly to symptomatic atherosclerosis and to disease progression. In the study, we use residual material from angioplasty catheter balloons and from vascular surgery plus blood samples. It is the hypothesis that material left on the catheter balloons used for angioplasty can be used for proteomics and metabolomics evaluation that will identify inflammation-associated proteins and signaling pathways directly in the diseased vessel. The tissue samples will be collected after the procedure and blood samples will be collected at the procedure plus after 6-12 months. The tissue and blood samples will be analyzed using mass spectrometry methods and a standard panel of biomarkers will also be analyzed using standardized methods. The analyses will include study of inflammation-associated peptides observed in autoinflammation as well as thrombogenic signaling pathways and local expression of biomarkers. The analyses of proteins, metabolites and/or biomarkers will be compared between cases (stable angina, unstable angina/non-STEMI, STEMI and vascular surgery) and controls (procedures not related to coronary artery diseases) to identify molecular processes related directly to symptomatic atherosclerosis and will be associated with disease progression using data from medical journals and National Health registries. The study will recruit 225 patients from Rigshospitalet University Hospital, Copenhagen, and Herlev-Gentofte Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atherosclerotic disease
* 18 years or older
* Angioplasty or vascular surgery

Exclusion Criteria:

- Not willing or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have their angioplasty or vascular surgery at the Copenhagen University hospital (Rigshospitalet) or Herlev-Gentofte hospital
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Protein composition in tissue | Baseline
  Difference in protein composition in tissue (residual material from angioplasty balloons) and blood samples compaired between study groups.
Metabolomic composition | Baseline
  Difference in metabolite composition in tissue (residual material from angioplasty balloons) and blood samples compaired between study groups.

SECONDARY OUTCOMES:
Biomarker composition | Baseline
  Differences in biomarker composition between groups
Biomarker composition | Within 12 months
  Differences in biomarker composition between groups
Disease progression in relation to protein, metabolite and biomarker compostion | With 12 months
  Changes in disease progression in relation to the protein, metabolite and biomarker composition
Disease progression in relation to protein, metabolite and biomarker compostion | 3 years
  Changes in disease progression in relation to the protein, metabolite and biomarker composition
Protein composition | Within 12 months
  Difference in protein composition in blood samples
Metabolomic composition | Within 12 months
  Difference in metabolite composition in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Gorm M Hansen, MD, PhD, Principal Investigator — The Heart Center, Rigshospitalet
Locations (2):
- Denmark (2):
  - The Heart Centre, Copenhagen
  - Herlev-Gentofte, Gentofte Municipality

IPD SHARING:
Plan to Share IPD: No